CLINICAL TRIAL: NCT02788175
Title: An Exploratory, Open-Label Study of Vedolizumab (Anti-alpha4beta7 Antibody) in Subjects With HIV Infection Undergoing Analytical Treatment Interruption
Brief Title: Vedolizumab (Anti-alpha4beta7) in Subjects With HIV Infection Undergoing Analytical Treatment Interruption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160118; 16-I-0118
Record Dates: First submitted 2016-05-28; First posted 2016-06-02 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2019-03-04

CONDITIONS: HIV
Keywords: HIV Immune Therapy; Monoclonal Antibody; Integrin
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIV-infected Adults on cART (Experimental): HIV-infected Adults (age 18 - 65) on CART with suppressed viremia
  Interventions: Biological: Entyvio (Vedolizumab)

INTERVENTIONS:
Biological: Entyvio (Vedolizumab) — A humanized monoclonal antibody that specifically binds to the alpha4beta7 integrin with MAdCAM-1, which in turn inhibits the migration of T-lymphocytes across the endothelium into GALT

SUMMARY:
Background:

In most people infected with human immunodeficiency virus (HIV), their immune system cannot control HIV infection. They need drugs called combination antiretroviral therapy (cART) to control the HIV. When people stop cART treatment, their immune system cannot control the infection again. They can also become resistant to cART and have lasting side effects. Researchers want to test if the drug vedolizumab is effective at controlling HIV infection without the need for cART.

Objective:

To test if vedolizumab is safe and can control the amount of HIV in the blood when cART is not taken.

Eligibility:

People ages 18-65 who have HIV and are being treated with cART

Design:

Participants will be screened with:

Physical exam

Medical history

Electrocardiogram: Soft, sticky patches on the chest, arms, and legs measure heart activity.

Blood and urine tests

Participants will have a baseline visit. This will be 2-5 hours each day for 1-2 days. It will include repeats of the screening tests and:

Leukapheresis: Blood is removed through a needle in the arm. A machine separates the white blood cells from the blood. The rest of the blood is returned to the participant.

Neurologic exam: The nerves and reflexes are tested.

First vedolizumab infusion through an arm vein

Participants will have visits every 4 weeks for 30 weeks. These will include:

Vedolizumab infusions

Repeats of baseline tests

Participants will have more visits for blood draws.

Participants will keep taking cART until after the week 22 infusion.

After discontinuing cART at study week 22, participants will be seen every two weeks to monitor the CD4 count and the level of HIV in the blood. Some of these visits will occur in between infusion visits and will only take about 1 hour to complete. cART will be restarted if a participant's HIV levels go up to high, or if their CD4 cell counts decreases by too much.

For the follow-up phase, participants will have visits every 4 weeks for 24 weeks. These will include blood tests and a physical exam.

...

DETAILED DESCRIPTION:
While combination antiretroviral therapy (cART) has improved the clinical outcome for HIV-infected individuals, persistence of viral reservoirs in the peripheral blood and lymphoid tissues remains a hurdle to complete eradication of virus and cure of the infection. The concept that HIV preferentially infects discrete subsets of CD4+ T cells underscores the need to develop therapeutics that exploit specific cell-virus interactions. T cells expressing integrin alpha4beta7 not only regulate migration into the gut associated lymphoid tissue (GALT), but also concomitantly bind HIV, placing them in a prime position to disseminate HIV throughout the tissue. Previously, it has been shown that the HIV envelope protein gp120 binds to alpha4beta7 on CD4+ T cells in vitro, alpha4beta7high CD4+ T cells are highly susceptible to productive HIV infection in vitro, and the administration of anti-alpha4beta7 monoclonal antibody (mAb) prevents and/or delays transmission of SIV upon repeated challenges and preserves CD4+ T cells in rhesus macaques. Furthermore, it has been demonstrated that administration of anti-alpha4beta7 mAb in SIV-infected rhesus macaques receiving cART suppresses plasma viremia for extended periods following discontinuation of cART, collectively suggesting that sustained virologic remission in the absence of cART may be achieved via direct targeting of alpha4beta7 integrin. It is well established that the vast majority of HIV-infected individuals treated with cART experience plasma viral rebound within weeks of cessation of therapy. Considering that current research on the treatment of HIV-infected individuals has been heavily focused on developing strategies aimed at achieving sustained virologic remission in the absence of cART, it is of great interest to investigate whether administration of anti-alpha4beta7 mAb can prevent plasma viral rebound and allow durable suppression of viral replication in HIV infected individuals after discontinuation of cART. We propose to examine the effect of vedolizumab, an FDA approved anti-alpha4beta7 mAb for the treatment of ulcerative colitis and Crohn's disease, on plasma viral rebound in HIV-infected individuals following analytical treatment interruption (ATI).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age, 18 - 65 years
2. Documented HIV-1 infection and clinically stable
3. In general good health, with an identified primary health care provider for medical management of HIV infection and willing to maintain a relationship with a primary health care provider for medical management of HIV infection while participating in the study
4. CD4+ T cell count >450 cells/mm3 at screening
5. Documentation of continuous cART treatment with suppression of plasma viral level below the limit of detection for more than or equal 2 years. Subjects with blips (i.e., detectable viral levels on cART) prior to screening may be included provided they satisfy the following criteria:

   1. The blips are <400 copies/mL, and
   2. Succeeding viral levels return to levels below the limit of detection on subsequent testing
6. Willingness to undergo ATI
7. Laboratory values within pre-defined limits at screening:

   * Absolute neutrophil count >1,000/mm3
   * Hemoglobin (Hgb) levels >10.0 g/dL for men and >9.0 g/dL for women
   * Platelet count >100,000/mm3
   * Prothrombin time (PT) and partial thromboplastin time (PTT) <1.5 upper limit of normal (ULN)
   * Estimated glomerular filtration rate (eGFR) of greater than or equal to 50 mL/min as determined by the NIH Clinical Center laboratory
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels of <1.1 x ULN. Total bilirubin <1.1 x ULN (unless subject is taking atazanavir or has Gilbert s Syndrome)
8. Willingness to have samples stored for future research

Participation of Women:

Contraception: The effects of vedolizumab on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

EXCLUSION CRITERIA:

1. Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen (HBsAg), or chronic hepatitis C virus (HCV) infection, as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
2. Documented nadir CD4+ T cell count <200 cells /mm3
3. Documented multiclass antiretroviral drug resistance that, in the judgment of the investigator, would pose a risk of virologic failure should additional mutations develop during the study
4. HIV immunotherapy or vaccine(s) received within 1 year prior to screening
5. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment
6. Receipt of other investigational study agent within 28 days of enrollment
7. Any active malignancy that may require systemic chemotherapy or radiation therapy
8. Systemic immunosuppressive medications received within 3 months prior to enrollment. The following are not excluded: [1] corticosteroid nasal spray or inhaler; [2] topical corticosteroids for mild, uncomplicated dermatitis; and [3] oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur (length of therapy less than or equal to 10 days, with completion in more than or equal to 30 days prior to enrollment)
9. History or other clinical evidence of:

   * Significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction)
   * Severe illness, chronic liver disease, malignancy, immunodeficiency other than HIV, active systemic infection other than HIV, or any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study
   * Active or latent tuberculosis, regardless of treatment history
10. Neurologic or neuropsychiatric disorder, the symptoms of which mimic PML and could interfere with the assessment of safety (e.g. history of encephalitis with motor sequela, stroke with sequela, severe major depressive disorder, severe bipolar disorder, seizure disorder)
11. Active drug or alcohol abuse or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements
12. Pregnancy or breast-feeding

Co-enrollment Guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies. Study staff should be notified of co-enrollment as it will require the approval of the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05-28; Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arthos J, Cicala C, Martinelli E, Macleod K, Van Ryk D, Wei D, Xiao Z, Veenstra TD, Conrad TP, Lempicki RA, McLaughlin S, Pascuccio M, Gopaul R, McNally J, Cruz CC, Censoplano N, Chung E, Reitano KN, Kottilil S, Goode DJ, Fauci AS. HIV-1 envelope protein binds to and signals through integrin alpha4beta7, the gut mucosal homing receptor for peripheral T cells. Nat Immunol. 2008 Mar;9(3):301-9. doi: 10.1038/ni1566. Epub 2008 Feb 10. PMID 18264102
- [Background] Cicala C, Martinelli E, McNally JP, Goode DJ, Gopaul R, Hiatt J, Jelicic K, Kottilil S, Macleod K, O'Shea A, Patel N, Van Ryk D, Wei D, Pascuccio M, Yi L, McKinnon L, Izulla P, Kimani J, Kaul R, Fauci AS, Arthos J. The integrin alpha4beta7 forms a complex with cell-surface CD4 and defines a T-cell subset that is highly susceptible to infection by HIV-1. Proc Natl Acad Sci U S A. 2009 Dec 8;106(49):20877-82. doi: 10.1073/pnas.0911796106. Epub 2009 Nov 20. PMID 19933330
- [Background] Byrareddy SN, Kallam B, Arthos J, Cicala C, Nawaz F, Hiatt J, Kersh EN, McNicholl JM, Hanson D, Reimann KA, Brameier M, Walter L, Rogers K, Mayne AE, Dunbar P, Villinger T, Little D, Parslow TG, Santangelo PJ, Villinger F, Fauci AS, Ansari AA. Targeting alpha4beta7 integrin reduces mucosal transmission of simian immunodeficiency virus and protects gut-associated lymphoid tissue from infection. Nat Med. 2014 Dec;20(12):1397-400. doi: 10.1038/nm.3715. Epub 2014 Nov 24. PMID 25419708

RESULTS

PARTICIPANT FLOW:
Groups:
- Vedolizumab in HIV-infected Adults on cART: HIV-infected Adults (age 18 - 65) on CART with suppressed viremia
Period: Overall Study
Arm/Group | Vedolizumab in HIV-infected Adults on cART
Started (Screened) | 26
Received Study Agent | 20
Completed | 13
Not Completed | 13
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible prior to study agent | 6

BASELINE CHARACTERISTICS:
Arm/Group | Vedolizumab in HIV-infected Adults on cART
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 15
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 2 or Higher Related Adverse Events
Description: The primary endpoint was the number of grade 2 or higher adverse events, including serious adverse events, that were probably or definitely related to vedolizumab.
Time Frame: From the start of the initial infusion until up to 72 weeks.
Population: The analyses included all subjects who received at least one infusion of vedolizumab
Measure: Number; unit: Events
Arm/Group | Vedolizumab in HIV-infected Adults on cART
Number analyzed (Participants) | 20
Events | 11

2. Secondary Outcome: Number of Subjects Who Met Criteria to Restart Antiretroviral Therapy Before Week 48
Description: The secondary endpoint was defined as number of subjects who experienced plasma viremia following ATI and met criteria to restart cART before week 48 [a confirmed >30% decline in baseline CD4+ T Cell count or an absolute CD4+ T Cell count in the setting of detectable HIV viremia (>40 copies/mL); a sustained (>4weeks) HIV RNA level of > 1000 copies/mL, or any HIV related symptoms or pregnancy.]
Time Frame: From Week 22 until up to 48 weeks.
Population: The analyses includes all subjects who entered into the analytical treatment interruption at Week 22
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab in HIV-infected Adults on cART
Number analyzed (Participants) | 18
Participants | 13

ADVERSE EVENTS:
Time Frame: up to 72 weeks
Arm/Group | Vedolizumab in HIV-infected Adults on cART
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab in HIV-infected Adults on cART (N=20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab in HIV-infected Adults on cART (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Campylobacter gastroenteritis (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Giardiasis (Infections and infestations) | 1
Gonorrhoea (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 8
Otitis media acute (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood bicarbonate decreased (Investigations) | 8
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 5
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 9
Blood magnesium decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 7
Blood potassium decreased (Investigations) | 3
Blood sodium decreased (Investigations) | 2
Blood sodium increased (Investigations) | 2
Eosinophil count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02788175/Prot_SAP_001.pdf